CLINICAL TRIAL: NCT06510803
Title: Sevoflurane Concentrations During Induction of Anesthesia With the Drager Apollo and GE Ohmeda Workstations in Children
Brief Title: Sevoflurane Concentrations in Children
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesia, State University of New York at Buffalo
Other Study IDs: 00008573
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Anesthetic; Sevoflurane; Age
Keywords: sevoflurane; anesthesia; children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Control is GE Ohmeda: The control group will utilize the GE Ohmeda workstation for induction of anesthesia with sevoflurane.
  Interventions: Drug: The case intervention is the sevoflurane concentrations with the Drager Apollo workstation

INTERVENTIONS:
Drug: The case intervention is the sevoflurane concentrations with the Drager Apollo workstation — The increases in the sevoflurane concentrations during induction of anesthesia with the Drager Apollo compared with the GE Ohmeda workstations

SUMMARY:
The sevoflurane concentrations (as well as vital signs, child's date of birth, type of surgery) will be recorded during the first 10 minutes of anesthesia.

DETAILED DESCRIPTION:
Protocol definition:

This study will not deviate from standard anesthetic management of children with the exception of recording the child's vital signs and anesthetic gas concentrations during the anesthetic induction.

Healthy children, 2-6 years of age, fasting and unmedicated scheduled to undergo minor elective surgery under general anesthesia at Oishei Children's Hospital in Buffalo, NY will be consented for this protocol by the principal investigator. Parents who speak English will be approached for consent; the formal hospital translator service will be used for those parents who do not speak English. The medical translator will translate the consent form for the parents.

Children will be selected for inclusion in this study from the elective surgery list. A total of 28 children of both sexes will be enrolled, 14 with each of the two workstations. We will strive to include the workstation in each operating room at least once in the study. The choice of anesthesia workstations, Drager Apollo or GE Ohmeda, is predetermined by the floor on which the surgery is planned. Drager Apollo workstations are deployed in each of the 7 pediatric operating rooms on the second floor at Oishei and GE Ohmeda workstations are deployed in each of the 5 pediatric operating rooms on the third floor at Oishei.

Once the standard anesthesia monitors are applied, the children will undergo a routine inhalational induction that begins with a mixture of 5 liters/minute nitrous oxide and 2 liters/minute oxygen. Once the end-tidal nitrous oxide concentration reaches 0.45, the sevoflurane vaporizer will be dialed to 8%. The inspired and expired concentrations of sevoflurane will be recorded at the designated times (see data collection sheet) for the first 10 minutes of anesthesia. All vital signs (oxygen saturation, end-tidal carbon dioxide tension, blood pressure and heart rate) will also be recorded.All unusual movements and airway responses will also be recorded and when they occurred (under Notes on the data collection form). At the conclusion of the 10 minutes of the induction, the airway will be secured with an airway device, the surgery will proceed as planned and the recording will cease. The study will be terminated.

The inspired and expired concentrations of Sevoflurane with the Drager Apollo and GE Ohmeda workstations over time will be summarized and displayed graphically. The maximum inspired concentrations of Sevoflurane during each induction with the two types of workstations will be compared using Student's t-test at a significance level of P<0.05.

Jerrold Lerman MD, FRCPC, FANZCA July 11, 2024

ELIGIBILITY:
Inclusion

* scheduled for elective surgery under general anesthesia,
* ASA physical status 1 or 2

Exclusion Criteria:

* parents refuse consent
* presence of moderate or severe cardiorespiratory disease
* difficult airway
* malignant hyperthermia
* neuromuscular disorders
* obesity
* obstructive sleep apnea

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children scheduled for ambulatory surgery at Oishei Children's Hospital in Buffalo on both the second and third floors of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Sevoflurane concentrations (inspired and expired concentrations) during induction of anesthesia | 10 minutes of induction of anesthesia
  We will measure the inspired and expired sevoflurane concentrations using an agent monitor during the first 10 minutes of induction

SECONDARY OUTCOMES:
Other effects | First 10 minutes of anesthesia
  all untoward events including airway responses, unexpected movements will be recorded
Maximum sevoflurane concentrations during induction of anesthesia | 10 minutes of induction of anesthesia
  The maximum sevoflurane concentrations (inspired and expired) during the first 10 minutes of induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, FRCPC, Principal Investigator — Great lakes anesthesiology
Locations (1):
- John R. Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
I am not interested in sharing the data.